CLINICAL TRIAL: NCT02033122
Title: Effect of Aerobic Training on Bronchial Hyperresponsiveness and Systemic Inflammation in Patients With Moderate or Severe Asthma: a Randomized Controlled Trial
Brief Title: Effect of Aerobic Training in Moderate or Severe Asthmatic Patients
Acronym: ETA1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigação em Imunologia (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETA1
Record Dates: First submitted 2013-10-31; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Asthma.
Keywords: exercise, bronchial hyperresponsiveness, inflammation
MeSH Terms: conditions — Asthma; Motor Activity; Bronchial Hyperreactivity; Inflammation | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic training (Active Comparator): the intervention will be an aerobic training program. For the TG subjects, breathing exercises will have duration of 30 minutes and will be always followed by aerobic training sessions that will consist in 35 minutes divided in 5 minutes of warm-up, 25 minutes of aerobic training and 5 minutes of cool down. Initially, aerobic training will be performed at the heart rate (HR) corresponding to one third of the difference between the anaerobic threshold (AnT) and the respiratory compensation point (RCP) obtained in the incremental cardiopulmonary testing (CPET) and after two weeks of the adaptation, the intensity will increased to two thirds of the difference between AnT and RCP. The program will be performed twice a week, for 3 months.
  Interventions: Other: Aerobic training; Other: Breathing exercise
- Breathing exercise (Sham Comparator): Patients from the control group will be taught breathing exercises with 30 min per session , twice a week , during 3 months. Every exercise will be performed in sets of 3 (2 min each) and 60 s of rest .
  Interventions: Other: Breathing exercise

INTERVENTIONS:
Other: Aerobic training — the intervention will be an aerobic training program. For the TG subjects, breathing exercises will have duration of 30 minutes and will be always followed by aerobic training sessions that will consist in 35 minutes divided in 5 minutes of warm-up, 25 minutes of aerobic training and 5 minutes of cool down. Initially, aerobic training will be performed at the heart rate (HR) corresponding to one third of the difference between the anaerobic threshold (AnT) and the respiratory compensation point (RCP) obtained in the incremental cardiopulmonary testing (CPET) and after two weeks of the adaptation, the intensity will increased to two thirds of the difference between AnT and RCP. The program will be performed twice a week, for 3 months.
  Arms: Aerobic training
Other: Breathing exercise — Patients from the control group will be taught breathing exercises with 30 min per session , twice a week , during 3 months. Every exercise will be performed in sets of 3 (2 min each) and 60 s of rest .

SUMMARY:
Exercise training has been proposed as adjunctive therapy in asthma to improve many clinical outcomes; however its effects on bronchial hyperresponsiveness (BHR) and inflammation, characteristic features in asthma, remains poorly understood. We aim to investigate the effects of aerobic training on BHR (primary aim) and systemic inflammation (secondary aim). In addition, clinical control and health related quality of life (HRQoL) will be also assessed.

DETAILED DESCRIPTION:
This is a randomized, controlled and single-blind trial whose intervention will be an aerobic training. Fifty -eight patients with moderate or severe persistent asthma will be recruited at a university hospital and randomly assigned in two groups: control (CG) or training (TG) .The study will be performed between two medical visits with intervals of six months and during this period the same medication dosage will be maintained. Patients in CG will perform (an educational program + breathing exercise; n=28) and TG patients will perform (an educational program+breathing exercises+aerobic training; n=30).The sessions will be conducted twice a week, for 3 months. Before and after the intervention, all patients will be evaluated by bronchial hyperresponsiveness, serum cytokines levels, total immunoglobulin E, induced sputum, fractional exhaled nitric oxide (FeNO), asthma clinical control (daily symptoms dairy, exacerbations and asthma control questionnaire - ACQ), health related quality of life (HRQoL); asthma quality of life questionnaire-(AQLQ), pulmonary function and cardiopulmonary exercise testing. All the patients will be evaluated by specific immunoglobulin E (atopy) through (skin prick test or Phadiatop).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate and severe persistent asthma
* Asthma will diagnosed according to Global Initiative for Asthma (GINA)
* Body Mass Index <35 kg/ m2
* Patients will submitted the medical treatment, followed by pulmonary specialists for at least 6 months.

Patients will considered clinically stable (i.e., no exacerbation or changes in medication for at least 30 days).

Exclusion Criteria:

* Patients will diagnosed with cardiovascular, musculoskeletal or other chronic lung diseases;
* Patients with current participation in exercise programs
* current smokers or ex-smokers will excluded from the study.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Bronchial hyperresponsiveness | Before and after 3 months of intervetion
  The bronchial provocation test will be conducted according to American Thoracic Society (ATS) guideline (1999). Patients will inhale increasing concentrations of histamine following the sequences: 0.0625, 0.25, 1.0, 4.0 and 16.0 mg/ ml using the method of the dosimeter (DeVilbiss 646nebulizer, DeVilbiss Health Care, USA) . Forced expiratory volume in one second (FEV1) will be measured after 30 and 90 seconds from the end of inhalations. The test will considered positive when the concentration of histamine promotes a fall ≥ 20% in FEV1 (PC20) with respect to the post-saline value or when the maximum concentration is reached (16 mg/mL).

SECONDARY OUTCOMES:
serum cytokines levels | Before and after 3 months of intervention
  The plasma levels of inflammatory mediators will be evaluated before and after 3 months of intervention.The method Cytometric Beat Array (CBA) (BD Biosciences, USA) will be used to analyze the levels of interleukins (IL) IL-4, IL-5, IL-6, IL-8, IL -10, Tumor Necrosis Factor (TNF-α) and IL-12p70 and chemokines IL-8, Monocyte Chemotactic Protein-1 (MCP-1/CCL2) and RANTES

OTHER OUTCOMES:
Clinical control | before and after 3 months of intervention
  Clinical control will be evaluated by daily symptoms dairy , exacerbation and asthma control questionnaire (ACQ) and
Health related quality of life | before and after 3 months of interventions
  Health related quality of life will be assessed by the Asthma Quality Life Questionnaire (AQLQ) .

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Giavina-Bianchi, MD, PhD, Principal Investigator — Univeristy of São Paulo
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, Brazil

REFERENCES:
- [Derived] Franca-Pinto A, Mendes FA, de Carvalho-Pinto RM, Agondi RC, Cukier A, Stelmach R, Saraiva-Romanholo BM, Kalil J, Martins MA, Giavina-Bianchi P, Carvalho CR. Aerobic training decreases bronchial hyperresponsiveness and systemic inflammation in patients with moderate or severe asthma: a randomised controlled trial. Thorax. 2015 Aug;70(8):732-9. doi: 10.1136/thoraxjnl-2014-206070. Epub 2015 Jun 10. PMID 26063507